CLINICAL TRIAL: NCT06847594
Title: Superhydration Versus Dextrose 10% for Prevention of Post Operative Nausea and Vomiting After Laparoscopic Cholecystectomy (prospective Randomised Controlled Study)
Brief Title: An Evaluation the Effect of Superhydration Versus Dextrose 10% for Prevention of Post Operative Nausea and Vomiting After Laparoscopic Cholecystectomy (prospective Randomised Controlled Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FMASU MS129/2024
Record Dates: First submitted 2025-01-15; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2024-12

CONDITIONS: Postoperative Nausea and Vomiting (PONV)
Keywords: postoperative nausea and vomiting; nausea; vomiting; laparoscopic cholecystectomy; superhydration; glucose 10%; dextrose 10%
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Nausea; Vomiting | interventions — Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Superhydration group receiving 20 ml/kg (Active Comparator): Group Ringer Lactate planned to receive ringer lactate 20 ml/kg over the first 90 to 120 minutes
  Interventions: Drug: ringer lactate (20ml/kg)
- Dextrose group receiving Dextrose 10% (Experimental): Group Dextrose planned to receive Dextrose 10% 250 ml over 60 minutes added to 3 ml/kg/Hr ringer lactate as intraoperative fluid maintenance
  Interventions: Drug: Dextrose 10%
- control group receiving 3ml/kg/hr (No Intervention): Group control planned to receive ringer lactate with rate 3ml /kg /Hr as intraoperative fluid maintenance added to the loading dose according to Ain Shams Anesthesia and Critical care department protocol

INTERVENTIONS:
Drug: ringer lactate (20ml/kg) — ringer lactate 20 ml/kg over the first 90 to 120 minutes after induction intraoperatively
  Other Names: Superhydration
  Arms: Superhydration group receiving 20 ml/kg
Drug: Dextrose 10% — Dextrose 10% 250 ml over 60 minutes
  Arms: Dextrose group receiving Dextrose 10%

SUMMARY:
The goal of this clinical trial is to learn if Dextrose 10% or superhydration works to prevent postoperative nausea and vomiting in patients undergoing laparoscopic cholecystectomy.

. The main questions it aims to answer are:

Does Dextrose 10% or superhydration lower the number of times participants gets an episode of nausea and vomititng after laparoscopic cholecystectomy surgery? Researchers will compare Dextrose 10% versus superhydration to a placebo (a look-alike substance that contains no drug) to see if glucose 10% or superhydation can work to prevent postoperative nausea and vomiting.

Participants will:

Take Dextrose 10% or superhydration or a placebo in the operation monitored for 4 hours after surgery to check on their nausea and vomiting state

ELIGIBILITY:
Inclusion Criteria:

1. Age: 21- 60 years
2. Patients with ASA classification I and II

Exclusion Criteria:

1. Declining to give written informed consent.
2. Patients with morbid obesity (BMI > 40).
3. ASA classification III-V.
4. Sever hypertension and heart failure.
5. Significant hepatic or renal disorder.
6. Patients with diagnosed diabetes mellitus type 1 or type 2.
7. Patients with history of PONV currently receiving steroids or antiemetics.
8. Pregnant or menstruating patients.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 204 (Actual)
Dates: Start 2024-02-25 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
To compare the incidence of Post operative nausea and vomiting in the study treatment groups | Postoperative 4 hours stay in PACU

SECONDARY OUTCOMES:
Frequency of vomiting episodes | Postoperative 4 hours stay in PACU
Measurement of PONV severity scores | Postoperative 4 hours stay in PACU
  Severity of PONV was assessed using a 4-point Verbal Descriptive Scale (VDS) which consists of:
  Score 0= no PONV: no complaint of nausea or vomiting; Score 1= mild PONV: patient complains from nausea but doesn't need antiemetic treatment.
  Score 2= moderate PONV: patient complains from nausea and need antiemetic treatment; Score 3= severe PONV: patient complains from nausea with episode of vomiting requiring antiemetic treatment.
  PONV scores were obtained every half hour
Time from extubation till discharge from PACU | From the moment of extubation till the moment of discharge from PACU with patient being completely vitally stable and nausea and vomiting free , assessed to be from 4 to 8 hours
total antiemetic medication consumption | Postoperative period 4 hours stay in PACU. ( if the patient needed to stay for longer duration in the PACU for any medical reason then any antiemetic used in this period will be recorded as well )
  Severity of PONV was assessed using a 4-point Verbal Descriptive Scale (VDS) which consists of:
  Score 0= no PONV: no complaint of nausea or vomiting; Score 1= mild PONV: patient complains from nausea but doesn't need antiemetic treatment.
  Score 2= moderate PONV: patient complains from nausea and need antiemetic treatment; Score 3= severe PONV: patient complains from nausea with episode of vomiting requiring antiemetic treatment.
  PONV scores were obtained every half hour, Rescue antiemetic granisetron 1 mg IV was given when VDS scores were 2 or more. Medications were given only after excluding other causes of PONV such as hypovolemia, hypotension, hypoxia. The total number of doses of antiemetics used were obtained every half hour from the time of entry to the PACU for 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Aya H. M. Ahmad, Assistant professor, MD, Principal Investigator — Ain Shams University Faculty of Medicine; Wael A. M. Abdelwahab, Assistant professor, MD, Principal Investigator — Ain Shams University Faculty of Medicine; Mohamed A. Elgendy, Assistant professor, MD, Study Director — Ain Shams University Faculty of Medicine
Locations (1):
- Faculty of Medicine Ain Shams University, Cairo, Abbassia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The IPD that will be shared will be Age, Sex, BMI, ASA score , operation duration and anesthesia duration , PONV severity score, nausea and vomiting frequency , total antiemetic usage intra and postoperative in the PACU and time needed to discharge from the PACU
Supporting Information: Study Protocol, CSR

REFERENCES:
- [Background] Stephenson SJ, Jiwanmall M, Cherian NE, Kamakshi S, Williams A. Reduction in post-operative nausea and vomiting (PONV) by preoperative risk stratification and adherence to a standardized anti emetic prophylaxis protocol in the day-care surgical population. J Family Med Prim Care. 2021 Feb;10(2):865-870. doi: 10.4103/jfmpc.jfmpc_1692_20. Epub 2021 Feb 27. PMID 34041090